CLINICAL TRIAL: NCT02949349
Title: Mycophenolate Mofetil Versus Azathioprine for Maintenance Therapy of Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBL15-001
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Lupus Nephritis
Keywords: Systemic Lupus Erythematosus; Lupus Nephritis; Mycophenolate Mofetil; Azathioprine; Maintenance Therapy; Prednisolone; Serum albumin; Serum creatinine; Spot urine protein/creatinine ratio
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — Mycophenolic Acid; Azathioprine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MMF 500mg (Experimental): Mycophenolate mofetil 500mg, PO BID
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisolone
- MMF 750mg (Experimental): Mycophenolate mofetil 750mg, PO BID
  Interventions: Drug: Mycophenolate mofetil; Drug: Prednisolone
- AZA (Active Comparator): Azathioprine 1mg/kg, PO BID
  Interventions: Drug: Azathioprine; Drug: Prednisolone

INTERVENTIONS:
Drug: Mycophenolate mofetil — Provided as 250mg/capsule, dose specific for each arm, orally twice a day, for 24 weeks.
  Other Names: Mycocep Capsules
  Arms: MMF 500mg; MMF 750mg
Drug: Azathioprine — Provided as 50mg/tablet, 1mg/kg, orally twice a day, for 24 weeks.
  Other Names: Imuran Azathioprine Tablets
  Arms: AZA
Drug: Prednisolone — Daily dose not more than 10mg, orally, for 24 weeks.

SUMMARY:
This study is designed to compare the safety and efficacy of Mycocep Capsules (Mycophenolate Mofetil) and a marketed Azathioprine formulation, Imuran Azathioprine Tablets, in the maintenance therapy of lupus nephritis.

DETAILED DESCRIPTION:
This study is designed to compare the two different doses of Mycocep Capsules (1.0g/day & 1.5g/day) and Imuran Azathioprine Tablets (2mg/kg/day), all in combination with low-dose prednisolone (≤10mg/day) as maintenance treatment for lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lupus nephritis.
* Currently receiving maintenance therapy with Azathioprine, Mycophenolate Mofetil, Mycophenolate Sodium, or Cyclosporine for lupus nephritis for at least 3 months prior to randomization.
* Stable use of low dose (≤10mg/day) oral prednisolone for lupus nephritis for at least 3 months prior to randomization.

Exclusion Criteria:

* Untreated, not in need of immunosuppressive treatment (in addition to corticosteroids), currently receiving induction therapy, or not responding to Azathioprine, Mycophenolate Mofetil or Mycophenolate Sodium as induction or maintenance therapy for lupus nephritis.
* Currently receiving or anticipated to receive cyclophosphamide or IV pulse of corticosteroids.
* Currently receiving continuous dialysis starting more than 2 weeks before randomization, and/or with an anticipated duration of more than 8 weeks.
* Previous kidney transplant or planned transplant.
* Presence of life threatening complications such as cerebral lupus or severe infection.
* Presence of liver dysfunction.
* Presence of COPD or asthma requiring oral steroids.
* Presence of bone marrow insufficiency or pure red cell aplasia unrelated to active systemic lupus erythematosus.
* Presence of persistent hematuria or pyuria for causes other than lupus nephritis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Change in serum albumin | 24 weeks treatment
Change in serum creatinine | 24 weeks treatment
Change in spot urine protein/creatinine ratio | 24 weeks treatment

SECONDARY OUTCOMES:
Change in serum albumin | 12 weeks treatment
Change in serum creatinine | 12 weeks treatment
Change in spot urine protein/creatinine ratio | 12 weeks treatment
Change in cholesterol | 24 weeks treatment
Change in triglyceride | 24 weeks treatment
Change in complete blood count/differential count (CBC/DC) | 24 weeks treatment
Change in number of subjects with doubling of serum creatinine | 24 weeks treatment
Change in the average daily dose of oral prednisolone | 24 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Han Chen, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan, R.O.C.

IPD SHARING:
Plan to Share IPD: No